CLINICAL TRIAL: NCT03624309
Title: Anlotinib Plus Docetaxel Versus Docetaxel for Treatment of EGFR Wild-type Advanced Non-small-cell Lung Cancer After Disease Progression on Platinum-based Therapy : a Multicentre, Double-blind, Randomised Explorative Trial
Brief Title: Anlotinib Plus Docetaxel for the Treatment of EGFR Wild-type Advanced Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry); Hunan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Wu, Chief director of department, Hunan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L018
Record Dates: First submitted 2018-08-05; First posted 2018-08-10 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib Plus Docetaxel (Experimental): Anlotinib (12mg QD PO d1-14, 21 days per cycle) and Docetaxel (75mg/m2 IV d1)
  Interventions: Drug: Anlotinib Plus Docetaxel
- Docetaxel (Active Comparator): Docetaxel (75mg/m2 IV d1)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Anlotinib Plus Docetaxel — Anlotinib (12mg QD PO d1-14, 21 days per cycle) and Docetaxel (75mg/m2 IV d1)
  Other Names: Anlotinib & Docetaxel
  Arms: Anlotinib Plus Docetaxel
Drug: Docetaxel — Docetaxel (75mg/m2 IV d1)
  Arms: Docetaxel

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase Ⅲ study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Therefore,we envisage using anlotinib plus docetaxel treat the EGFR wild-type advanced Non-small cell lung cancer patients who were failure in the treatment of chemotherapy with platinum containing drugs, to further improve the patient's PFS or OS.

DETAILED DESCRIPTION:
This is a multicentre randomised controlled clinical trial conducted in China to compare the effectiveness and safety of Anlotinib Plus Docetaxel in patients of EGFR wild-type Advanced Non-squamous Non-small Cell Lung Cancer.

Eligible patients will be randomized to arm A and arm B:

Arm A: Patients on the anlotinib and docetaxel arm received 75mg/m2 docetaxel as intravenous infusion on day 1 of a 21-day cycle and 12mg anlotinib orally daily on day 1to 14 of a 21-day cycle.

Arm B: Patients on the docetaxel arm received 75mg/m2 docetaxel as intravenous infusion on day 1 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* diagnosed with advanced NSCLC (phase IIIB/IIIC/IV) through pathology, with measurable nidus(using RECIST 1.1)
* have failed for platinum two drugs chemotherapy
* EGFR wild type
* ECOG PS：0-1,Expected Survival Time: Over 3 months
* main organs function is normal
* the woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 2 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 2 months after it

Exclusion Criteria:

* Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer)
* have used docetaxel before
* have used antiangiogenic drugs （except Bevacizumab or endostatin）
* have failed for two times or beyond of platinum two drugs chemotherapy（except adjunctive therapy，neoadjuvant therapy and concurrent chemoradiotherapy ）
* iconography (CT or MRI) shows that the tumor vessels have 5 mm or less, or Cardiovascular involvement by Central tumor ; Or obvious lung empty or necrotic tumor
* patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination revealed brain or leptomeningeal disease） (28 days before the random treatment has been completed and the symptoms of patients with brain metastases from stable can into the group, but need to the cerebral MRI, CT or vein angiography confirmed as without symptoms of cerebral hemorrhage)
* patients are participating in other clinical studies (other than non-interventional studies) less than 4 weeks from the end of a previous clinical study
* other kinds of malignancies within 5 years or for now
* have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
* abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or be treated with thrombolysis and anticoagulation
* urine routines show urine protein≥ ++, or urine protein quantity≥ 1.0 g during 24 hours
* uncontrollable hypertensive (systolic blood pressure or greater 150 mmHg or diastolic blood pressure or greater 90 mmHg, despite the best drug treatment)
* the effects of surgery or trauma had been eliminated for less than 14 days before admission to the study group
* patients with severe infections , and need to receive Systemic antibiotic treatment
* significant cardiac disease as defined as: grade II or greater myocardial infarction, unstable arrhythmia(Including corrected QT interval (QTc )period between male or greater 450 ms, female or greater 470 ms); New York Heart Association (NYHA) grade II or greater heart dysfunction , or Echocardiography reveal left ventricular ejection fraction （LVEF）Less than 50%
* patients with NCI-CTCAE grade II or greater peripheral neuropathy, except due to trauma
* pleural effusion or ascites, resulting in respiratory syndrome (≥CTC AE level 2)
* serious, non-healing wound, ulcer, or bone fracture
* decompensated diabetes or high dose glucocorticoid treatment of other contraindication
* has an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* has Clinically significant hemoptysis Within 3 months before Random (daily hemoptysis than 50 ml;Or significant clinical significance of bleeding symptoms or have definite bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers, baseline period + + and above of fecal occult blood, or vasculitis, etc
* has venous thromboembolism events Within 12 months before Random, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc
* whole body antitumor treatment was planned in the first 4 weeks(except diphosphonate) or during this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy， Chinese medicine with antitumor effect. Field scale radiotherapy (EF-RT) within 4 weeks before grouping or limited field radiotherapy before grouping were carried out in 6 months ;
* a known history of HIV testing positive or acquired immunodeficiency syndrome (AIDS)
* untreated active hepatitis (hepatitis b: HBsAg positive and HBV DNA more than 1 x 103 copy /ml; Hepatitis c: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection
* serious diseases that endanger patients' safety or affect patients' completion of research,according to the researchers' judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | each 42 days up to PD or death(up to 24 months)
  Progress free survival

SECONDARY OUTCOMES:
OS | From randomization until death (up to 24 months)
  Overall Survival
ORR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate
DCR | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate
Safety (Number of Participants with Adverse Events as a Measure of Safety and Tolerability) | Until 21 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: LIN WU, professor, Principal Investigator — Hunan cancer hospital,Tongzipo Road 283#, Hunan,China
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Pu X, Shou J, Xiao Z, Chen J, Xiao M, Guo Q, Ma Z, Hong W, Wang Q, Wang Y, Li J, Rao C, Weng J, Lu L, Wu L, Fang Y. Anlotinib Plus Docetaxel is Promising in Advanced NSCLC Progressing on First-Line Immunotherapy: A Pooled Analysis of Two Randomized Trials. Adv Ther. 2025 Jul;42(7):3249-3264. doi: 10.1007/s12325-025-03170-2. Epub 2025 May 12. PMID 40354010